CLINICAL TRIAL: NCT04407442
Title: Phase II Study of Daratumumab in Combination With Azacitidine and Dexamethasone in Relapsed/Refractory Multiple Myeloma Patients Previously Treated With Daratumumab
Brief Title: Daratumumab, Azacitidine, and Dexamethasone for Treatment of Patients With Recurrent or Refractory Multiple Myeloma Previously Treated With Daratumumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment and change in sponsor direction
Sponsor: University of California, San Francisco (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20251; NCI-2020-02985 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-05-22; First posted 2020-05-29 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Azacitidine; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (azacitidine, dexamethasone, daratumumab) (Experimental): PRE-INDUCTION (CYCLE 0): Patients receive azacitidine IV on days -7 to -3 in absence of disease progression or unacceptable toxicity.
  INDUCTION (CYCLES 1-2): Patients receive azacitidine IV on days 22-26, dexamethasone IV or orally (PO), and daratumumab subcutaneously (SC) over 3-5 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity
  CONSOLIDATION (CYCLES 3-6): Patients receive azacitidine IV on days 22-26 of cycle 3 and on days 1-5 of cycles 5-6, dexamethasone IV or PO, and daratumumab SC over 3-5 minutes on days 1 and 15. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity
  MAINTENANCE (CYCLES 7+): Patients receive azacitidine IV on days 1-5, dexamethasone IV or PO, and daratumumab SC over 3-5 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Azacitidine; Biological: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Biological: Daratumumab — Given SC
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex

SUMMARY:
This phase II trial studies how well daratumumab, azacitidine, and dexamethasone work in treating patients with multiple myeloma that has come back (recurrent) or has not responded to treatment (refractory) and was previously treated with daratumumab. Daratumumab is an antibody made up of immune cells that attaches to a protein on myeloma cells, called cluster of differentiation 38 (CD38). CD38 is found in higher levels on tumor cells than on normal cells. Daratumumab prevents the growth of tumors who have high levels of CD38 by causing those cells to die. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dexamethasone is a steroid that helps decrease inflammation and lowers the body's normal immune response to help reduce the effect of any infusion-related reactions. Giving azacitidine may help increase the levels of CD38 on the tumor cells to increase the function of daratumumab to attach to those tumor cells to help destroy them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of adding azacitidine to daratumumab and dexamethasone, as measured by the overall response rate in patients with relapsed refractory multiple myeloma (RRMM) previously treated with daratumumab.

SECONDARY OBJECTIVES:

I. To evaluate the duration of response per International Myeloma Working Group (IMWG) criteria.

II. To evaluate the safety and tolerability of azacitidine in combination with daratumumab and dexamethasone.

III. To evaluate progression free and overall survival in patients treated with azacitidine in combination with daratumumab and dexamethasone.

IV. To assess the changes in CD38 expression on plasma cells after treatment with azacitidine and correlate this change with the depth and duration of response of azacitidine in combination with daratumumab and dexamethasone.

OUTLINE:

PRE-INDUCTION (CYCLE 0): Patients receive azacitidine intravenously (IV) on days -7 to -3 in the absence of disease progression or unacceptable toxicity.

INDUCTION PHASE (CYCLES 1-2): Patients receive azacitidine IV on days 22-26 and dexamethasone IV or orally (PO) and daratumumab subcutaneously (SC) over 3-5 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION PHASE (CYCLES 3-6): Patients receive azacitidine IV on days 22-26 of cycle 3 and on days 1-5 of cycles 5-6 and dexamethasone IV or PO and daratumumab SC over 3-5 minutes on days 1 and 15. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE (CYCLES 7+): Patients receive azacitidine IV on days 1-5 and dexamethasone IV or PO and daratumumab SC over 3-5 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. Patients must have a known diagnosis of multiple myeloma with evidence of measurable disease, AND have evidence of disease progression based on IMWG criteria:

   * Serum M-protein >= 0.5 g/dL, or urine M-protein >= 200 mg/24 hours. OR
   * In the absence of measurable M-protein, serum immunoglobulin free light chain >= 10 mg/dL, and abnormal serum immunoglobulin kappa lambda free light chain ratio
3. Relapsed from or refractory to 2 or more different prior therapies, including immunomodulatory drugs (IMiDs; e.g., thalidomide, lenalidomide) and proteasome inhibitors, chemotherapy-based regimens, monoclonal antibodies, or autologous stem cell transplantation (ASCT)

   * Relapse is defined as progression of disease after an initial response (minimal response (MR) or better) to previous treatment, more than 60 days after cessation of treatment
   * Refractory disease is defined as < 25% reduction in M-protein or progression of disease during treatment or within 60 days after cessation of treatment
4. Prior exposure to daratumumab, with most recent dose being at least 6 months prior to trial enrollment
5. Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%)
6. Demonstrates adequate organ function as defined below within 7 days of first dose of drug:

   * Absolute neutrophil count >= 1,500/microliter (mcL)
   * Platelets >= 75,000/mcL
   * Total bilirubin within normal institutional limits, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits
   * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) =< 3 x institutional upper limit of normal
   * Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 3 x institutional upper limit of normal
   * Creatinine =< 1.5 x within institutional upper limit or normal OR creatinine clearance glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation, unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
7. Life expectancy of at least 3 months
8. Women of childbearing potential must have at least one negative highly sensitive serum (beta-human chorionic gonadotropin (beta-hCG)) during screening, within one week prior to the first dose of any component of study treatment
9. Before enrollment, a woman must be either:

   * Not of childbearing potential defined as:

     * Postmenopausal:

       * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone level (> 40 IU/L or milli-international units per milliliter (mIU/mL) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy, however in the absence of 12 months of amenorrhea, a single follicle stimulating hormone measurement is insufficient
     * Permanently sterile

       * Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy OR
   * Of childbearing potential and

     * Practicing 2 highly effective user-independent methods of contraception (failure rate of < 1% per year when used consistently and correctly

       * Examples of highly effective user-independent methods of contraception include:

         * Implantable progesterone-only hormone contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); vasectomized partner; sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the subject.)
       * Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical studies
       * Hormonal contraception may be susceptible to interaction with the study drug, which may reduce the efficacy of the contraceptive method
       * Agrees to remain on a highly effective method for 4 weeks before the first dose of any component of study treatment, throughout the study (including during dose interruptions), and for 4 weeks following discontinuation of azacitidine, and for 3 months after last daratumumab dose

         * Note: If the risk of pregnancy changes (e.g., a woman who is not heterosexually active becomes active), a woman must begin a highly effective method of contraception, as described throughout the inclusion criteria

           * If reproductive status is questionable, additional evaluation should be considered
       * Agrees to not breast feed for the duration of the study (including during dose interruptions), and for 4 weeks following discontinuation of azacitidine, and for 3 months after last daratumumab dose
10. Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study (including during dose interruptions), and for 4 weeks following discontinuation of azacitidine, and if receiving daratumumab, for 3 months after the last dose
11. Due to the teratogenicity of azacitidine and the lack of adequate reproductive toxicity data for daratumumab, in addition to the user independent highly effective method of contraception, a male or female condom with or without spermicide, diaphragm, or cervical cap is required. Male condom and female condom should not be used together (due to risk of failure with friction)
12. During the study (including during dose interruptions), and for 4 weeks following discontinuation of azacitidine, and for 3 months after the last daratumumab dose, in addition to the user independent highly effective method of contraception (even if he has undergone a successful vasectomy), a man

    * Who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (i.e., latex or synthetic condom with spermicidal foam/gel/film/cream/suppository)
    * Who is sexually active with a woman who is pregnant must use a latex or synthetic condom
    * Must agree not to donate sperm
13. Willing and able to adhere to the prohibitions and restrictions specified in this protocol and referenced in the informed consent form (ICF)
14. Must sign an ICF (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

1. Diagnosed or treated for malignancy (either solid tumor or hematologic) other than multiple myeloma, except:

   * Malignancy treated with curative intent and with no known active disease before enrollment

     * Adequately treated non-melanoma skin cancer, lentigo maligna or in situ malignancies (including but not limited to, cervical, breast) with no evidence of disease
2. Received daratumumab therapy less than 6 months prior to trial enrollment
3. Primary refractory to prior daratumumab
4. Subject is:

   * Seropositive for human immunodeficiency virus (HIV)
   * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen (anti-HBc) and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
   * Seropositive for hepatitis C (except in the setting of a sustained virologic response (SVR), defined as aviremia at least 12 weeks after completion of antiviral therapy)
5. Known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal to minimize daratumumab-related pulmonary toxicities

   * Note: FEV1 testing is required for subjects suspected of having chronic obstructive pulmonary disease and asthma. Subjects must be excluded if FEV1 < 50% of predicted normal
6. Known moderate or severe persistent asthma within the past 2 year or currently has uncontrolled asthma of any classification

   * Note: Subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study. FEV1 testing is required for subjects suspected of having asthma
7. Concurrent medical condition or disease (e.g., active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study
8. Clinically significant cardiac disease, including:

   * Myocardial infarction within 6 months before cycle 1, day -7, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association class III-IV)
   * Uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities
   * Screening 12-lead electrocardiogram (ECG) showing a baseline corrected QT interval (QTc) > 470 msec.
9. Known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, daratumumab or its excipients (refer to investigator's brochure), or known sensitivity to mammalian-derived products
10. Concurrent plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and/or skin changes), or light chain amyloidosis
11. Known or suspected of not being able to comply with the study protocol (e.g., because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments
12. Contraindications to the use of daratumumab, azacitidine or dexamethasone per local prescribing information
13. Taken any disallowed therapies before the planned first dose of study drug
14. Received any therapy to treat cancer (including radiation, chemotherapy, biologics, cellular therapies, and/or steroids at doses > 20 mg) or undergone a major surgical procedure within 14 days, or within 5 half-lives of an anticancer drug, prior to the first dose of study treatment, whichever is longer (with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma).
15. Participated in an interventional clinical trial(s) and received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before cycle 1, day -7 or 5 pharmacokinetic half-lives, whichever is longer.
16. Had major surgery within 2 weeks before cycle 1, day -7, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study or within 2 weeks after the last dose of study drug administration. Note: Subjects with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty is not considered a major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Chung, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  60-69 years old | 3
  70-79 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants with either a stringent complete response (sCR) + complete response (CR) + very good partial response + partial response (PR) as best response using International Myeloma Working Group (IMWG) Uniform Response Criteria for all subjects who have measurable disease and received at least 2 cycles of study treatment, and have at least 2 efficacy evaluation assessments.
Time Frame: Up to 18 months
Population: One participant has insufficient imaging data required for efficacy evaluation and was excluded from this analysis
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 4
proportion of participants | 0.75

2. Secondary Outcome: Number of Participants With Reported Treatment-related Adverse Events (AE)
Description: All safety analyses for AEs will be based on all subjects who receive at least 1 cycle of study treatment. AEs will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 from the initiation of study treatment until discontinuation of treatment. For each treatment-related adverse event, the number of subjects who experience at least 1 occurrence of the given event which was attributed to the study regimen as probable, possible or definite will be summarized.
Time Frame: Up to 18 months
Measure: Number; unit: participants
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 5
participants
  Injection site reaction | 4
  White blood cell decreased | 1
  Chills | 1
  Hyperglycemia | 1
  Insomnia | 1
  Diarrhea | 1
  Lymphocyte count decreased | 1
  Nausea | 2
  Platelet count decreased | 1
  Pruritus | 1
  Sore Throat | 1
  Upper respiratory infection | 1
  Eye Pain | 1
  Neutrophil count decreased | 3

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease according to the IMWG criteria or death due to progressive disease whichever occurred first all subjects who have measurable disease and received at least 2 cycles of study treatment, and have at least 2 efficacy evaluation assessments. DOR will be summarized using the Kaplan-Meier estimator. Median even-free survival will be reported and the corresponding 95% confidence interval will be calculated using Brookmeyer and Crowley method.
Time Frame: Up to 18 months
Population: One participant has insufficient imaging data required for efficacy evaluation and was excluded from this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 4
months | 9.1 [1.4 to NA] — There were insufficient number of events so an upper limit could not be calculated

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the date of first dose of study treatment to the date of death due to any cause or censored based on the date of last encounter if patient is alive or lost to follow-up. OS will be summarized using the Kaplan-Meier estimator. Median even-free survival will be reported and the corresponding 95% confidence interval will be calculated using Brookmeyer and Crowley method.
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 5
months | NA [10.1 to NA] — There were insufficient number of events (N=1) to determine median OS and upper limit of confidence interval could not be calculated

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the date of first dose of study treatment to the date of first documented evidence of progressive disease or death, whichever occurs first. PFS will be summarized using the Kaplan-Meier estimator. Median even-free survival will be reported and the corresponding 95% confidence interval will be calculated using Brookmeyer and Crowley method.
Time Frame: Up to 18 months
Population: One participant has insufficient imaging data required for efficacy evaluation and was excluded from this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 4
months | 10.3 [2.66 to NA] — There were insufficient number of events so an upper limit could not be calculated

6. Secondary Outcome: Change in CD38 Surface Expression of Plasma Cells
Description: Change in CD38 surface expression will be summarized using descriptive statistics and tested using the one-sample t-test. Two-sided p-value less than 0.05 will be considered statistically significant.
Time Frame: Starting 6 days before treatment up until the end of cycle 1 (each cycle is 28 days); up to 34 days total
Population: Data not collected for this endpoint
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Patients Who Achieve at Least 1.5 Fold Increase in Their CD38 Expression
Description: Will be assessed by flow cytometry and based on a one-sample t-test at a two-sided type I error rate of 0.05.
Time Frame: At the end of cycle 1 (each cycle is 28 days)
Population: Data not collected for this endpoint
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 0

8. Secondary Outcome: Correlation of Change in CD38 Expression After Azacitidine With Overall Response
Description: Will be correlated to overall response using logistic regression, linear regression methods, and Spearman's correlation coefficient, as appropriate.
Time Frame: Up to 18 months
Population: Data not collected for this endpoint
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 0

9. Secondary Outcome: Correlation of Change in CD38 Expression After Azacitidine Treatment With Depth of Response
Description: Correlation will be calculated using logistic regression, linear regression methods, and Spearman's correlation coefficient, as appropriate.
Time Frame: Up to 18 months
Population: Data not collected for this endpoint
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 0

10. Secondary Outcome: Correlation of Change in CD38 Expression After Azacitidine With Duration of Response
Description: Will be correlated to duration of response using logistic regression, linear regression methods, and Spearman's correlation coefficient, as appropriate.
Time Frame: Up to 18 months
Population: Data not collected for this endpoint
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Treatment (Azacitidine, Dexamethasone, Daratumumab)
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine, Dexamethasone, Daratumumab) (N=5)
Upper respiratory infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine, Dexamethasone, Daratumumab) (N=5)
Fever (General disorders) | 4 (5)
Injection site reaction (General disorders) | 4 (13)
Fatigue (General disorders) | 3 (6)
Chills (General disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (13)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (4)
White blood cell decreased (Investigations) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Penile infection (Infections and infestations) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed to enrollment earlier than expected due to slow enrollment and change in sponsor research direction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT04407442/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT04407442/ICF_001.pdf